CLINICAL TRIAL: NCT03912571
Title: Sleep Disordered Breathing and Alzheimer's Disease Biomarkers in Normal Aging and Mild Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12-00041
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mild Cognitive Impairment (MCI): Patients with clinical dementia rating of 0.5 or a global deterioration scale of 3.
  Interventions: Diagnostic Test: Structural 3T MRI; Diagnostic Test: MRI Based Perfusion Imaging; Diagnostic Test: VR-CO2 MRI Scans
- Normal Cognition (NL): Clinical Dementia Rating [CDR] of 0 or Global Deterioration Scale [GDS] of 1-2
  Interventions: Diagnostic Test: Structural 3T MRI; Diagnostic Test: MRI Based Perfusion Imaging; Diagnostic Test: VR-CO2 MRI Scans

INTERVENTIONS:
Diagnostic Test: Structural 3T MRI — measures of global and hippocampal atrophy)
Diagnostic Test: MRI Based Perfusion Imaging — brain blood flow
Diagnostic Test: VR-CO2 MRI Scans — reduced vaso reactivity to carbon dioxide

SUMMARY:
The purpose of this study is to determine the sleep patterns of subjects with or without sleep disturbances (insomnia, sleep apnea) and compare these findings with their previous FDG/PIB PET, structural MRI and brain blood flow scams performed during their participation in the Following studies 'Alzheimer's Disease Core Center (ADCC) Clinical Evaluation' (IRB: 2942), MRI Progression Markers of Cognitive Decline in the Elderly' (IRB:09-0586), or 'Imaging Neuro inflammation in Alzheimer's Disease with [11C] Arachidonic Acid (AA) and PET'(IRB: 10-00442).

ELIGIBILITY:
Inclusion Criteria:

* All subjects will have participated in prior CBH studies and have agreed to an FDG, PIB and MRI scans.

Exclusion Criteria:

* Diagnosis of sleep apnea and under treatment with a continuous positive airway pressure (CPAP) machine.
* Active depressive episode during the evaluation with a Geriatric Depression Scale score >7 and/or a Clinical Global Impression scale for depression score >4.
* Moderate Cognitive decline (GDS >3).
* Severe primary or secondary insomnia except insomnia due to SDB.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 cognitively healthy subjects (normal or MCI) previously enrolled in Alzheimer's Disease Core Center (ADCC) and CBH studies who have agreed to be contacted about future research studies will be asked to additionally participate in this study. The age range of the subjects will be of 55-90 years based on the incidence of dementia in middle age and elder adults.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-11-13 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Decreased cerebral blood flow (CBF) | 1 Week
  Measured by perfusion MRI
Measure of vasoreactivity to CO2 (VRCO2) | 1 Week
  subjects will breath through a respiratory tube and CO2 will be meaured
Increase in cortical AB plaque burden | 1 Week
  Measured by PIB PET

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Osorio, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Medical Center, New York, New York, United States